CLINICAL TRIAL: NCT03852459
Title: A Randomized, Double-Blind,Vehicle-Controlled Study to Determine the Efficacy and Safety of AP0302 in the Treatment of Delayed Onset Muscle Soreness (DOMS)
Brief Title: Controlled Study to Assess the Efficacy and Safety of S-Ibuprofen Topical Gel 5% (AP0302) in the Treatment of DOMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aponia Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-007
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-05

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: active gel and matching vehicle control gel
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): S-Ibuprofen Topical Gel 5%
  Interventions: Drug: S-Ibuprofen
- Placebo Arm (Placebo Comparator): Vehicle Topical Gel
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: S-Ibuprofen — Topical Gel 5%
  Arms: Active Arm
Drug: Vehicle — Vehicle Gel
  Arms: Placebo Arm

SUMMARY:
Phase 2 study designed to evaluated analgesic efficacy and safety of S-Ibuprofen Topical Gel 5%

DETAILED DESCRIPTION:
The purpose of this randomized, double-blind study is to evaluate the efficacy and safety of S-Ibuprofen Topical Gel 5% in reducing pain/soreness associated with delayed onset muscle soreness (DOMS).

ELIGIBILITY:
Inclusion Criteria:

* history of pain/soreness after exercise
* BMI between 18-30
* negative drug, alcohol, pregnancy screens
* other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* upper extremity workout in last 3 months
* job or hobby requiring heavy lifting
* history of muscle disorders
* allergy or intolerance to NSAID or study drug
* history of recent pain medication use
* other protocol-defined exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 251 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, MD, Principal Investigator — JBR Research
Locations (1):
- JBR Clinical Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2/3, single-center study conducted in USA
Pre-assignment Details: A total of 434 subjects were screened in the study of which 251 subjects were randomized.
Groups:
- Active Arm: S-Ibuprofen Topical Gel 5%
  AP0302 (S-ibuprofen topical gel 5%)applied up to 7 times in 24 hours, over a 48-hour dosing period.
- Placebo Arm: Vehicle Topical Gel
  Placebo topical gel 5% applied up to 7 times in 24 hours, over a 48-hour dosing period.
Period: Overall Study
Arm/Group | Active Arm | Placebo Arm
Started | 126 | 125
Completed | 123 | 122
Not Completed | 3 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm | Placebo Arm | Total
Number analyzed (Participants) | 126 | 125 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (10.41) | 30.6 (10.37) | 29.4 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 68 | 141
  Male | 53 | 57 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 24 | 48
  Not Hispanic or Latino | 102 | 101 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 2 | 3
  White | 102 | 102 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 9 | 25
Region of Enrollment [Number; unit: participants]
  United States | 126 | 125 | 251
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.01 (3.146) | 24.55 (3.082) | 24.28 (3.120)

OUTCOME MEASURES:

1. Primary Outcome: Sum of the Time-weighted Differences From Baseline in Pain Intensity With Movement(SPIDMOVE) Over 24 Hours Post Time Zero
Description: The primary efficacy outcome is the sum of the time-weighted differences from baseline in muscle pain/soreness with movement over 0-24 hours post T0 (SPIDMOVE 0-24h), that is the area under the differences from baseline pain/soreness intensity difference curve. The pain intensity differences (PIDs) with movement from time point A to time point B was calculated using the trapezoid rule by subtracting each post-T0 pain score with movement from the pain score with movement at time point Ti. Positive and higher scores indicate greater reduction in pain. Measured by Pain Intensity Numerical Rating Scale (PI-NRS) where 0 = no pain and 10 = worst possible pain at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 26, 28, 30, 32, 34, 36, 40, 44, and 48 hours post-initial IP dose and immediately prior to the subsequent doses of investigational product (IP).
Time Frame: 0-24 hours.
Population: Full Analysis Set: All subjects who were randomized, received at least 1 dose of study drug, and had at least 1 post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 125
score on a scale*hours | -33.09 (31.311) | -29.09 (29.763)
Statistical Analysis 1: Comparison: Active Arm vs Placebo Arm; Test type: Superiority; p = 0.4272, ANCOVA

2. Secondary Outcome: SPIDMOVE Over the Following Intervals: 0-6, 6-12, 0-12, 12-24, 24-36, 24-48, 0-36, 36-48 and 0-48 Hours Post-T0.
Description: Sum of the time-weighted differences from baseline in pain intensity with movement (SPIDMOVE) over the following intervals: 0-6, 6-12, 0-12, 12-24, 24-36, 0-36, 24-28, 36-48, and 0-48 hours post-T0, that is the area under the differences from baseline pain/soreness intensity difference curve. The PIDs with movement from time point A to time point B was calculated using the trapezoid rule by subtracting each post-T0 pain score with movement from the pain score with movement at time point Ti. Positive and higher scores indicate greater reduction in pain. Measured by Pain Intensity Numerical Rating Scale (PI-NRS) where 0 = no pain and 10 = worst possible pain at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 26, 28, 30, 32, 34, 36, 40, 44, and 48 hours post-initial IP dose and immediately prior to the subsequent doses of IP.
Time Frame: From 0-6, 6-12, 0-12, 12-24, 24-36, 0-36, 24-28,36-48, and 0-48 hours post-T0. Time point i included 1, 2, 3, 4, 5, 6 (pre-dose), 7, 8, 9, 10, 11, 12 (pre-dose), 16, 18 (pre-dose), 20, and 24 (pre-dose) hours after the first dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 125
score on a scale*hours
  0-6 hours | -4.82 (5.478) | -4.06 (5.807)
  6-12 hours | -8.98 (8.583) | -7.73 (8.412)
  0-12 hours | -13.80 (13.435) | -11.79 (13.682)
  12-24 hours | -19.29 (18.868) | -17.30 (17.338)
  24-36 hours | -26.55 (18.582) | -24.35 (18.807)
  24-48 hours | -60.37 (38.168) | -54.61 (38.604)
  0-36 hours | -59.64 (48.384) | -53.44 (46.530)
  36-48 hours | -33.82 (20.293) | -30.26 (20.794)
  0-48 hours | -93.47 (66.331) | -83.71 (64.201)

3. Secondary Outcome: Sum of Time Weighted Differences From Baseline in Muscle Stiffness (SSID) With Movement Over the Interval
Description: Sum of the time-weighted differences from baseline in muscle stiffness with movement (SSIDMOVE) over the following intervals: 0-6, 6-12, 0-12, 12-24, 0-24, 24-36, 24-48, 0-36, 36-48, and 0-48 hours post-T0, that is the area under the differences from baseline stiffness difference curve. The muscle Stiffness Intensity Differences (SIDs) with movement from time point A to time point B was calculated using the trapezoid rule by subtracting each post-T0 stiffness score with movement from the stiffness score with movement at time point Ti. Positive and higher scores indicate greater reduction in stiffness. Measured by Muscle Stiffness Numerical Rating Scale (NRS) where 0 = No Stiffness and 10 = Worst Possible Stiffness at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 16, 20, 24, 26, 28, 30, 32, 34, 36, 40, 44, and 48 hours post-initial IP dose and immediately prior to the subsequent doses of IP.
Time Frame: 0-6, 6-12, 0-12, 12-24, 24-36, 24-48, 0-36, 36-48, and 0-48 post T0
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 125
score on a scale*hours
  0-6 hours | -3.81 (6.218) | -3.33 (5.957)
  6-12 hours | -7.75 (9.893) | -6.48 (8.796)
  0-12 hours | -11.55 (15.446) | -9.81 (14.302)
  12-24 hours | -17.20 (20.476) | -14.91 (19.369)
  0-24 hours | -28.75 (34.920) | -24.72 (32.365)
  24-36 hours | -23.33 (21.209) | -19.95 (22.555)
  24-48 hours | -53.58 (44.528) | -44.77 (44.732)
  0-36 hours | -52.08 (54.840) | -44.68 (53.031)
  36-48 hours | -30.25 (23.947) | -24.82 (23.171)
  0-48 hours | -82.33 (76.936) | -69.49 (73.804)

4. Secondary Outcome: Total Relief With Movement (TOTPAR) 0-6 Hours Post Time Zero
Description: Total relief with movement (TOTPAR) 0-6 hours post time zero
  TOTPAR was calculated as the sum of pain relief at time point i (PR i) times the weight for each PR i, where i referred to each pain relief scheduled assessment time point between A and B (not including B). The higher the number the better pain relief.
  Categorical Relief Rating Scale: Subjects rated relief from starting pain with movement using a 5-point categorical relief scale "0=no relief," "1=a little relief," "2=some relief," "3=a lot of relief," or "4=complete relief" at 1, 2, 3, 4, 5, and 6 hours post-initial IP dose and immediately prior to a subsequent dose of IP if one occurred prior to 6 hours.
Time Frame: 0-6 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale*hours
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 125
score on a scale*hours | 4.06 (3.435) | 3.61 (3.978)

5. Secondary Outcome: Subject Global Assessment of Study Medication Assessed at Approximately 48 Hours Post Time Zero
Description: Global assessment of efficacy will be assessed at approximately 48 hours post-T0 (or upon early termination if the subject withdraws prior to the 48-hour assessment).
  Subject Global Assessment Using Original 5 Categories as 0=poor, 1=fair, 2=good, 3=very good, 4=excellent. In addition, the 5 categories were dichotomized into 2 categories (good/very good/excellent versus poor/fair). The proportion of good, very good, and excellent ratings were calculated for each treatment.
Time Frame: 48 hours post time zero
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 124
Participants
  Original Categories - Poor | 44 | 50
  Original Categories - Fair | 48 | 47
  Original Categories - Good | 25 | 21
  Original Categories - Very good | 9 | 5
  Original Categories - Excellent | 0 | 1
  Dichotomized Categories - Poor/fair | 92 | 97
  Dichotomized Categories - Good/very good/excellent | 34 | 27

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAE was defined as an adverse event that was new or worsened in severity after the first dose of study drug. A treatment-related TEAE was defined as a TEAE that was at least possibly related to the administration of study drug or was missing the relationship assessment. If a TEAE was recorded on multiple occasions, only the highest severity was presented.
Time Frame: Up to Day 7
Population: Safety Population: All subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Active Arm | Placebo Arm
Number analyzed (Participants) | 126 | 125
participants
  Subjects with any TEAE | 125 | 121
  Subjects with any treatment-related TEAEs | 124 | 120
  Subjects with TEAEs leading to discontinuation | 2 | 2
  Subjects with SAEs | 0 | 0
  TEAE with mild in severity | 119 | 115
  TEAE with moderate in severity | 6 | 4
  TEAE with Severe in severity | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to Day 7
Description: TEAE was defined as an adverse event that was new or worsened in severity after the first dose of study drug.
Arm/Group | Active Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/125
Other Adverse Events (participants affected / at risk) | 123/126 | 117/125
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Arm (N=126) | Placebo Arm (N=125)
application site erythema (General disorders) | 123 | 117
application site induration (General disorders) | 25 | 21
application site pain (General disorders) | 70 | 13
application site pruritus (General disorders) | 62 | 76
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 8 | 8
skin exfoliation (Skin and subcutaneous tissue disorders) | 27 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT03852459/Prot_SAP_001.pdf